CLINICAL TRIAL: NCT05476523
Title: Development and Validation of a Novel Eye-Tracking Software-based Platform to Extract Oculometric Measures
Status: Recruiting | Type: Observational
Sponsor: NeuraLight (Industry)
Responsible Party: Sponsor
Other Study IDs: HDC/2022-3
Record Dates: First submitted 2022-07-25; First posted 2022-07-27 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Eye Movement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Data Collection: As a part of the study, a group of up to 2000 healthy subjects will undergo a NeuraLight session including oculometric measurements and eye-tracking recordings using a novel software-based platform and an eye-tracking system (approx. 15 minutes). The oculometric evaluation will occur for every patient 1 time, and all subjects will be recruited over a period of 36 months. All assessments will be performed during a clinic visit unless authorized to be conducted remotely
  Interventions: Other: NeuraLight

INTERVENTIONS:
Other: NeuraLight — NeuraLight is an investigational software-based platform used for measuring eye movements in response to visual stimuli and captured using a simple webcam

SUMMARY:
This is an observational prospective study in a cohort of healthy subjects who are enrolled using convenience and snowballing sampling. The aims of the study is to demonstrate the efficacy of using NeuraLight system to capture oculometric data from healthy participants and to validate the data capture of NeuraLight oculometric measurements as compared with a validated eye-tracker system in subjects who meet the inclusion criteria and who provide a signed Informed Consent.

DETAILED DESCRIPTION:
The purpose of the trial is to demonstrate the efficacy of using NeuraLight system to capture oculometric data from healthy participants, and to validate the data capture of NeuraLight oculometric measurements as compared with a validated eye-tracker system. In addition, we also aim to collect oculometric data from healthy participants in order to optimize a regression model which can be used for future prediction of clinical endpoints in various neurological patients at different stages of disease

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages between 18 and 90 years old
* Normal or corrected vision
* Ability to follow instructions
* Willing and able to sign an informed consent form

Exclusion Criteria:

* Inability to sit for 20 minutes on a chair in a calm manner
* Personal or 1st degree relative history of epilepsy
* Additional neurological diseases
* Drug or alcohol abuse

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy subjects
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-07-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of data capture | 36 months
  Capturing >50 different oculometric measures in >95% of a cohort of up to 2000 subjects
Validation of data capture | 36 months
  Relative root mean square error (RMSE) of NeuraLight's extracted oculometric measures compared with retrieved measurements from a validated eye tracking system <0.1

SECONDARY OUTCOMES:
Optimization of data capture | 36 months
  Optimization of a feature selection model (Fisher's Linear Discriminant Analysis (LDA)) on NeuraLight oculometric measures used for a logistic regression model of clinical endpoints with a relative root mean square error (RMSE) of <0.1

CONTACTS AND LOCATIONS:
Overall Officials: Eitan Raveh, PhD, Principal Investigator — NeuraLight
Locations (1):
- NeuraLight, Wilmington, Delaware, United States

IPD SHARING:
Plan to Share IPD: No